CLINICAL TRIAL: NCT01464996
Title: Clinical Evaluation Of A New Two-Component Self-Etch Universal Adhesive (OptiBond XTR)
Brief Title: Clinical Evaluation Of A New Two-Component Self-Etch Universal Adhesive
Acronym: XTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kerr Corporation (Industry)
Responsible Party: Principal Investigator, André V. Ritter, DDS, MS, Professor UNC School of Dentistry, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Kerr-XTR-11
Record Dates: First submitted 2011-10-25; First posted 2011-11-04 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Composite Restorations; Tooth Lesions
Keywords: non-carious cervical lesions; bonded restorations; composites; adhesives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adhesive OptiBond XTR (Experimental): Adhesive OptiBond XTR will include composite restorations placed using the dental adhesive OptiBond XTR.
  Interventions: Procedure: Adhesive: OptiBond XTR; Composite: Herculite Ultra
- Adhesive OptiBond FL (Active Comparator): Adhesive OptiBond FL will include composite restorations placed using the dental adhesive OptiBond FL.
  Interventions: Procedure: Adhesive: OptiBond FL; Composite: Herculite Ultra

INTERVENTIONS:
Procedure: Adhesive: OptiBond XTR; Composite: Herculite Ultra — The intervention in Arm 1 (Adhesive: OptiBond XTR; Composite: Herculite Ultra) is a 2-step, self-etching adhesive.
  Arms: Adhesive OptiBond XTR
Procedure: Adhesive: OptiBond FL; Composite: Herculite Ultra — Arm 2 (Adhesive: OptiBond FL; Composite: Herculite Ultra) is a 3-step, etch-and-rinse adhesive.
  Arms: Adhesive OptiBond FL

SUMMARY:
This randomized clinical trial evaluates the clinical performance of a new two-component self-etch universal adhesive, OptiBond XTR, when applied in non-carious Class V cervical lesions without macromechanical retention (retentive grooves or bevels). The control material is OptiBond FL, a "traditional" etch/prime/bond adhesive with documented clinical performance. Eighty non-carious Class V cervical lesions are divided into two groups to be treated with either OptiBond XTR or OptiBond FL. Both adhesives are applied strictly according to the manufacturer's directions. Herculite Ultra, a nano-hybrid resin-based composite, is used as the restorative material with both adhesives. The restorations will be evaluated at insertion (baseline), 6 months, and 18 months. An optional three-year recall evaluation is also proposed. The investigators hypothesize that both adhesives will have comparable performance.

DETAILED DESCRIPTION:
CLINICAL RESEARCH PLAN

Introduction

This randomized clinical trial involved the restoration and evaluation of 83 (target enrollment was 80) non-carious cervical lesions (NCCLs) using either the new two-component self-etch universal adhesive OptiBond XTR or a control dental adhesive, OptiBond FL, and a nano-hybrid composite restorative material, Herculite Ultra. OptiBond XTR is a two-component self-etch, filled, fluoride releasing, light-cured bonding agent designed for the universal bonding of direct and indirect restorations. The study design was based on the American Dental Association Acceptance Program Guidelines for Dentin and Enamel Adhesive Materials.

Participant Selection Criteria

Participants were selected on the basis of requiring restorations of non-carious cervical lesions. Participants with fewer than 20 teeth were not considered. The participant pool was randomized as much as possible to exclude bias due to age (18 to 80 years old), sex, race, national origin, or other factors such as unusual dietary, habitual, or oral hygiene factors which might affect the results. If the participant pool included these effects, they will be acknowledged in all project reports. Despite our efforts to have close to equal numbers of men and women in the study (ADA Guidelines, 2001), as noted in this report our pool was imbalanced towards women (we enrolled 20 females and 4 males). However, we do not believe this gender imbalance will affect or bias the results.

Prior to enrollment in the study, participants signed a consent form. Both the consent form and this research protocol were reviewed and approved by an Institutional Review Board (IRB) at the University of North Carolina. IRB approval was secured throughout the study.

Tooth Selection Criteria

Any tooth included in the study contacted the opposing tooth in a normal occlusal relationship and had normal periodontal health. The dental health status of the participant was considered normal in all respects except for ongoing restorative procedures in unrelated and unopposed quadrants.

Teeth restored had non-carious cervical lesions (NCCLs, abrasion/erosion/abfraction) with no undercuts. Class V carious lesions were excluded. Normally, no more than 50% of the cavosurface margin involved enamel and more than 75% of the surface area of the defect involved dentin.

All NCCLs were characterized preoperatively relative to height of the lesion, width, depth, percent of margin in enamel, internal angle of the lesion, and degree of sclerosis as measured by the UNC Sclerosis Scale (Appendix 1). The shape of the lesions was documented as "saucer-shaped" or "notch-shaped." Evidence of stressful occlusion (wear facets, fremitus) also was noted. These clinical co-variables can retrospectively be analyzed if any retention failures occur to assess potential cause and effect relationships.

Distribution of Restorations (Per Participant)

To minimize the chance that strong participant-related effects could distort the outcome of the study, no more than two restorations of each type of material (four total restorations) per participant were allowed. Our initial target was for the distribution of restorations to include approximately one-half anterior teeth and one-half posterior teeth. A minimum of 25 participants at baseline, 20 participants at 6 months, and 15 participants at 18 months is required for evaluation (ADA Guidelines, 2001).

A randomized schedule was prepared to minimize the effects of operator, participant, and material on the results of the study.

Participants were scheduled as they were accepted in the study, and operators were scheduled to place the restorations according to the Department of Operative Dentistry master schedule. For each participant, the adhesive used (OptiBond XTR or OptiBond FL) in the first restoration placed was chosen on the flip of a coin, and the subsequent restorations (if more than one tooth was to be restored on that participant) were done using the other adhesive and so on. Consequently, if the participant had two or more lesions to be restored, he/she received both adhesives. Every effort was made to distribute the restorations evenly in the mouth, i.e., restorations placed with both adhesives were equally distributed in anterior/posterior teeth, and in maxillary/mandibular teeth.

Tooth Preparation Procedures

All tooth preparations were of a modified design (as described in Sturdevant's Art and Science of Operative Dentistry, 6th edition, 2012). The preparations did not include retentive grooves or bevels. The dentin and enamel walls of the preparation were lightly roughened with a coarse diamond stone. Tooth preparation were limited to roughening the involved surfaces and producing a definite finish line, where indicated.

Operative procedures were performed using local anesthesia as needed. The operating sites were isolated with cotton rolls and retraction cord, or rubber dam, depending on access and location of the lesion.

Tooth Restoration Procedures

OptiBond XTR and OptiBond FL were applied according to the specific directions supplied by the manufacturer. The preparations were restored with a light-cured nanoparticle resin-based composite material (Herculite Ultra). The composite was inserted in increments of 2 mm or less. Each increment was fully polymerized according to composite shade for no less than 20 seconds using a Demi Plus LED light-curing unit as determined and provided by the manufacturer.

After polymerization, finishing was accomplished with 12-fluted tapered and/or flame-shaped carbide finishing burs using light intermittent pressure to avoid damaging the margins. Polishing was accomplished with slow speed polishing brushes (Occlubrush, Axis Dental) and aluminum-oxide polishing discs (OptiDisc, Axis Dental) where accessible.

Records

There are many factors that might contribute to retention and/or microleakage failures. For that reason, the following items were recorded on the project data forms (see Appendix 3 for example of data form) for each restoration placed during the course of the study:

1. Identification # of the operator
2. Tooth # for each restoration
3. Participant's age and gender for each restoration
4. Isolation method (e.g., cotton roll, retraction cord, rubber dam)
5. Number of increments of restorative composite
6. Shade of composite
7. Total polymerization time for adhesive and composite
8. Finishing technique and instruments used
9. Any unusual step and/or event (e.g., contamination requiring additional etching and/or application of adhesive)

Standardization of Clinicians (Operators)

This study was conducted with four operators experienced in this trial design. For the purpose of initial standardization, all project personnel met to review the procedures in detail, comparing their individual assessments of the procedures. They discussed difficulties and potential problems and finalized the details of all clinical procedures. All involved operators are full-time faculty of the Department of Operative Dentistry with years of experience in clinical research.

During the course of the insertions, the patient coordinator had primary responsibility for continual assessment of standardization. Any procedural step that was out of the ordinary was recorded on the project data forms (comments section) and signed. In addition, the principal investigators reviewed those points at the periodic meetings of the project personnel.

CLINICAL EVALUATION PLAN

Clinical Evaluation Times

The restorations were evaluated at insertion (baseline) and 6 months, and will be evaluated at 18 months, with an optional three-year evaluation. This document reports on data collected at the 6 month evaluation visit.

Direct Evaluation Criteria and Procedures

Each restoration will be evaluated for the following characteristics:

1. Retention
2. Color match
3. Cavosurface margin discoloration
4. Secondary caries
5. Anatomic form
6. Marginal adaptation and/or integrity
7. Post operative sensitivity

United States Public Health Service (USPHS) direct evaluation procedures will be conducted using the methods reported by Ryge in 1973. See Appendix 2 for a complete description of the Direct Evaluation Criteria. Retention will be recorded as completely retained (alfa) or partially or completely lost (charlie).

All restorations will be evaluated independently by two operators. Consensus will be determined by consultation and re evaluation. The individual and consensus values will be recorded on data sheets. The consensus values for each participant at baseline and each recall period will be recorded on a participant case card. The case card data will be transferred directly to a summary sheet containing data for all participants treated.

Indirect Evaluation Criteria and Procedures

Intraoral photographs are the best method to document color matching, interfacial staining, and occlusal patterns. Intraoral color photographs were taken at baseline (before and after restoration placement) and will be taken at each evaluation appointment as a permanent record for subsequent indirect evaluation and later reference. Pre-operative photographs consist of one image of the defect to be restored. Clinical photographs will be high-quality digital images made at an original magnification of 1.5x and will be used principally for reference to document the direct evaluations.

STATISTICAL ANALYSIS

Experimental Questions

This study will evaluate the retention and other aspects of a new two-component self-etch adhesive system in non-retentive cervical defects when compared to a resin adhesive system with documented performance. The study is designed so that its results can be compared with the results of previous clinical trials and with ADA guidelines.

Experimental Design

This randomized clinical trial is designed as an equivalence trial, i.e., the overall hypothesis tested is that the clinical performance of OptiBond XRT, as measured by the USPHS criteria described, will be equivalent to that of OptiBond FL, which has excellent documented clinical performance. In order to minimize possible participant and operator effects on the results of the study, the assignment of participants to operators and materials to teeth was randomized (see section Distribution of Restorations per Participant above). Participants were assigned to operators in order of screening.

Data Analysis

Individual clinical evaluations and consensus values shall be recorded at each recall visit and signed by each evaluator. Categorical (USPHS) values will be tabulated and incidence values will be reported for comparison to the specification limits. Any failures during the clinical study will be counted as failures in all subsequent recalls. The restorations' failure rates will be calculated using the following equation:

Failure Percentage = [(PF+NF)/(PF+RR)] x 100%

PF = Number of previous failures before the current recall NF = Number of new failures during the current recall RR = Number of restorations recalled for the current recall

Because the study is designed as an equivalence trial, the power calculation is based not on expected differences between adhesive systems, but rather on differences in performance of the systems across time (baseline versus evaluation times). For an estimated 30 percent difference in clinically unacceptable scores between baseline and 3 years, the sample size used will adequately power the study at 85 percent. At baseline, data on subjects' age, sex and occlusion, lesion characteristics and operator may be compared between the two restorative systems using two-sample t tests (continuous variables) and χ2 (categorical variables), to determine if the two groups are equivalent. The lesion characteristics to be evaluated are internal angle, percentage of enamel margin, sclerosis scale value, and lesion size (height, width and depth) and volume. Modified USPHS direct evaluation criteria scores of restorations placed with OptiBond XTR or OptiBond FL will be compared at each evaluation time for statistically significant differences using the Fisher exact test (P = 0.05). Lesions/restorations will be used as the unit of analysis (cases). Although restorations placed in the same participant are not totally independent cases, the assignment of restorations to participants was randomized. Therefore, subject and lesion characteristics are not expected to affect outcomes. However, to test for the influence of such characteristics on the performance of the restorative systems, logistic regression can be used to control for factors such as operator; subject's age, sex and occlusion; and lesion's location, size and score on the sclerosis scale. Finally, we will run a survival analysis and derive a Kaplan-Meier survival estimate curve on the clinically unacceptable (Charlie) scores for any of the USPHS criteria at the different follow-up times. A log rank test for equality of survivor function will be used to compare the survival estimates of the two restorative systems. We will use Stata 10 data analysis and statistical software (StataCorp, College Station, Texas) for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects needing restoration of NCCLs (these include some cases where the patient has hypersensitivity and a restoration is indicated)
* Subjects with age range 18-80 years old
* Teeth with normal occlusion relationships

Exclusion Criteria:

* Subjects with fewer than 20 teeth
* Subjects with poor oral hygiene and/or uncontrolled periodontal disease
* Teeth with NCCLs with mechanical undercuts
* Subjects with known allergies to HEMA or resin-based materials. The materials to be used are HEMA and/or resin-based materials.
* Subjects with medical conditions that contraindicate dental treatment.
* Subjects with xerostomia. Xerostomia is a condition where there is a decrease salivary flow (dry mouth). Decrease salivary flow is a known factor that affects the long-term prognosis of dental restorations, and would be a confounder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: André V Ritter, DDS, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill School of Dentistry, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty six participants were screened and satisfied inclusion criteria, but only 24 were enrolled.
Groups:
- All Study Participants: Will include composite restorations placed using both the dental adhesive OptiBond XTR and OptiBond FL.
  Participants were randomized to receive either type of intervention
Period: Overall Study
Arm/Group | All Study Participants
Started | 24
OptiBond XTR | 23
OptiBond FL | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: There were 24 participants in the study. The 24 participants received 83 restorations. As per protocol, participants received restorations from both arms, hence total number of study participants should not be the sum of the number of participants for each arm.
Groups:
- All Study Participants: Will include composite restorations placed using both dental adhesives OptiBond XTR and OptiBond FL.
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 4
Number of Restorations, Categorical [Number; unit: number of restorations, unit]
  OptiBond XTR | 41
  OptiBond FL | 42
Stressful Occlusion, Categorical [Number; unit: Number of teeth with stressful occlusion]
  OptiBond XTR | 20
  OptiBond FL | 20

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Overall retention of restorations
Time Frame: 6 and 18 months post-baseline
Population: what is reported here is the retention rate using the restoration as the unit of analysis
Measure: Number; unit: percentage of restorations
Units Other Than Participants: restorations
Groups:
- Adhesive OptiBond XTR: will include composite restorations placed using the dental adhesive OptiBond XTR.
  Adhesives: OptiBond XTR Composite: Herculite Ultra: The intervention in Arm 1 (XTR) is a 2-step, self-etching adhesive.
- Adhesive OptiBond FL: will include composite restorations placed using the dental adhesive OptibOnd FL.
  Adhesives: OptiBond FL Composite: Herculite Ultra: Arm 2 (FL) is a 3-step, etch-and-rinse adhesive.
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Number analyzed (Participants) | 23 | 24
Number analyzed (restorations) | 41 | 42
percentage of restorations
  6 months | 100 | 100
  18 months | 100 | 97

2. Secondary Outcome: Color Match
Description: Percentage of restorations that scored alfa. Restoration matches adjacent tooth structure in color, shade and translucency.
Time Frame: 18 months post-baseline
Measure: Number; unit: % of restorations with alfa scores
Units Other Than Participants: restorations
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Number analyzed (Participants) | 23 | 24
Number analyzed (restorations) | 41 | 42
% of restorations with alfa scores | 89 | 76

3. Secondary Outcome: Cavosurface Margin Discoloration
Description: Percentage of restorations scoring alfa. No discoloration is present anywhere on the margin between the restoration and the tooth structure.
Time Frame: 18 months post-baseline
Measure: Number; unit: % of restorations with alfa scores
Units Other Than Participants: restorations
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Number analyzed (Participants) | 23 | 24
Number analyzed (restorations) | 41 | 42
% of restorations with alfa scores | 89 | 92

4. Secondary Outcome: Secondary Caries
Description: Percentage of restorations with alfa scores. Absence of caries is evidenced by softness, opacity, or etching at the margin of the restoration.
Time Frame: 18 months post-baseline
Measure: Number; unit: % of restorations with alfa scores
Units Other Than Participants: restorations
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Number analyzed (Participants) | 23 | 24
Number analyzed (restorations) | 41 | 42
% of restorations with alfa scores | 100 | 100

5. Secondary Outcome: Anatomic Form
Description: Percentage of restorations with alfa scores. Restoration is continuous with existing anatomic form.
Time Frame: 18 months post-baseline
Measure: Number; unit: % of restorations with alfa scores
Units Other Than Participants: restorations
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Number analyzed (Participants) | 23 | 24
Number analyzed (restorations) | 41 | 42
% of restorations with alfa scores | 97 | 92

6. Secondary Outcome: Marginal Adaptation and/or Integrity
Description: Percentage of restorations with alfa scores. No discoloration is present anywhere on the margin between the restoration and the tooth structure.
Time Frame: 18 months post-baseline
Measure: Number; unit: % of restorations with alfa scores
Units Other Than Participants: restorations
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Number analyzed (Participants) | 23 | 24
Number analyzed (restorations) | 41 | 42
% of restorations with alfa scores | 97 | 89

7. Secondary Outcome: Post Operative Sensitivity
Description: Percentage of restorations with alfa scores. No sensitivity.
Time Frame: 18 months post-baseline
Measure: Number; unit: % of restorations with alfa scores
Units Other Than Participants: re
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Number analyzed (Participants) | 23 | 24
Number analyzed (re) | 41 | 42
% of restorations with alfa scores | 100 | 100

ADVERSE EVENTS:
Arm/Group | Adhesive OptiBond XTR | Adhesive OptiBond FL
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No